CLINICAL TRIAL: NCT02266914
Title: Magnetic Resonance Elastography of Cardiac Transplant Rejection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard D. White, M.D.,, Professor and Chair, Department of Radiology, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013H0318
Record Dates: First submitted 2014-09-30; First posted 2014-10-17 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Acute Graft Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Patients who have received a cardiac transplant at The Ohio State University Ross Heart Hospital will undergo Magnetic Resonance Elastography (MRE) (using a Magnetic Resonance Elastography driver) within 24-48 hours of standard of care biopsy. Results of both will be compared to determine if MRE can successfully predict cardiac transplant rejection.
  Interventions: Device: Magnetic Resonance Elastography driver

INTERVENTIONS:
Device: Magnetic Resonance Elastography driver — A driver is required for MRE. The driver utilizes sound waves to produce vibrations. Images of these vibrations are captured with Magnetic Resonance scanner to produce images that indicate stiffness in an organ.
  Other Names: Siemens MRE Driver

SUMMARY:
Magnetic Resonance Elastography (MRE) for cardiac transplant patients.

DETAILED DESCRIPTION:
Patient will undergo MRE beginning 4-8 weeks post transplant, then with each scheduled cardiac biopsy through 7-8 months post transplant. Results of the MRE will be compared against results of the cardiac biopsy to determine if the non-invasive MRE can predict cardiac transplant rejection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have undergone cardiac transplantation at the Ohio State University Ross Heart Hospital.
* Patients must be able to lie flat on their back in the scanner for up to 60 minutes
* Patient must be able to hold their breath for up to 15 seconds at a time.

Exclusion Criteria:

* Patients who are claustrophobic
* Patients who are pregnant, due to potential risks to the fetus.
* Patients with any unapproved, non-MRI safe metal/devices in their bodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard White, MD, Principal Investigator — The Ohio State University Medical Center Dept. of Radiology
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 27, 2014 to December 7, 2014 (approximately 1 year) at The Ohio State University Wexner Medical Center.
Groups:
- Cardiac Transplant Patients: Patients who have received a cardiac transplant at The Ohio State University Ross Heart Hospital will undergo Magnetic Resonance Elastography (MRE) (using a Magnetic Resonance Elastography driver) within 24-48 hours of standard of care biopsy. Results of both will be compared to determine if MRE can successfully predict cardiac transplant rejection.
  Magnetic Resonance Elastography driver: A driver is required for MRE. The driver utilizes sound waves to produce vibrations. Images of these vibrations are captured with Magnetic Resonance scanner to produce images that indicate stiffness in an organ.
Period: Overall Study
Arm/Group | Cardiac Transplant Patients
Started | 9
Completed | 0
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Transplant Patients
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Stiffness With Magnetic Resonance Elastography (MRE)
Description: MRE scans will be performed within 24-48 hours of standard of care cardiac biopsies for patients who have undergone cardiac transplant at The Ohio State University Ross Heart Hospital. Stiffness results from the MRE will be compared to histopathology from the cardiac biopsy to determine if the completely non-invasive MRE can successfully predict transplant rejection.
Time Frame: 24-48 hours
Population: Data were not collected due to study termination.
Arm/Group | Cardiac Transplant Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | Cardiac Transplant Patients
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-02-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT02266914/Prot_SAP_000.pdf
  • Informed Consent Form (2014-01-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT02266914/ICF_001.pdf